CLINICAL TRIAL: NCT04620200
Title: Neo-adjuvant Nivolumab or Nivolumab With Ipilimumab in Advanced Cutaneous Squamous Cell Carcinoma Patients Prior to Standard of Care Surgery; the MATISSE Trial
Brief Title: Neo-adjuvant Nivolumab or Nivolumab With Ipilimumab in Advanced Cutaneous Squamous Cell Carcinoma Prior to Surgery
Acronym: MATISSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N20MAT
Record Dates: First submitted 2020-08-20; First posted 2020-11-06 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cutaneous Squamous Cell Carcinoma
Keywords: immunotherapy; neoadjuvant; nivolumab; ipilimumab
MeSH Terms: interventions — Nivolumab; Immunotherapy; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARM A (Experimental): 2 courses of nivolumab 3 mg/kg in week 0 and 2 prior to standard of care
  Interventions: Drug: Nivolumab
- ARM B (Experimental): 2 courses of nivolumab 3 mg/kg in week 0 and 2 plus 1 course of ipilimumab 1mg/kg in week 0 prior to standard of care
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — 3mg/kg
  Other Names: immunotherapy
Drug: Ipilimumab — 1mg/kg
  Other Names: immunotherapy
  Arms: ARM B

SUMMARY:
To determine the histopathological response rate to neo-adjuvant nivolumab and nivolumab plus ipilimumab at time of standard of care(surgery ± radiotherapy).in patients with cutaneous squamous cell carcinoma.

DETAILED DESCRIPTION:
This is an investigator-initiated randomized non-comparative phase II trial consisting of 40 patients with resectable stage III-IVa CSCC randomized 1:1 to ARM A: 2 courses of nivolumab 3 mg/kg in week 0 and 2, or ARM B: 2 courses of nivolumab 3 mg/kg in week 0 and 2 plus 1 course of ipilimumab 1mg/kg in week 0. Both treatment arms are neo-adjuvant and applied prior to standard of care (consisting of surgery at week 4 with or without adjuvant radiotherapy).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Patient is able to understand and comply with the protocol requirements and has signed the informed consent form.
3. World Health Organization (WHO) Performance Status 0 or 1 (Appendix B).
4. Patients with histologically or cytologically confirmed, primary or recurrent stage III-IVA CSCC of all body sites.

   OR

   Patients with histologically or cytologically proven stage I-II CSCC, only in the case of:
   * Presence of multifocal disease for which extensive and/or mutilating surgery is necessary (e.g. near-total scalp resection).
   * Situated in an anatomical localization that necessitates extensive and/or mutilating surgery (e.g. orbital exenteration).
5. Eligible for standard-of-care, curatively intended surgery with or without adjuvant radiotherapy.
6. Screening laboratory values must meet the following criteria: WBC ≥ 2.0x109 /L, Neutrophils ≥1.5x109 /L, Platelets ≥100 x109 /L, Hemoglobin ≥5.5 mmol/L, Creatinine ≤1.5x ULN, AST ≤ 1.5 x ULN, ALT ≤ 1.5 x ULN, Bilirubin ≤1.5 X ULN (except subjects with Gilbert Syndrome, who are eligible when total bilirubin < 3.0 mg/dL).
7. Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. They should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of the investigational drug.
8. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25IU/L or equivalent units of HCG) prior to the start of nivolumab or nivolumab + ipilimumab.
9. Men who are sexually active with WOCBP must use a contraceptive method with a failure rate of less than 1% per year and will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product. Surgically sterile or azoospermic men do not require aforementioned contraception.

Exclusion Criteria:

1. Distantly metastasized (stadium IVb) CSCC.
2. SCC localized in a mucosal surface (i.e. anus, vulva, penis or mucosal portion of lip).
3. Patients for whom SOC consists of definitive (brachy)radiotherapy.
4. Primary or recurrent CSCC appearing in an area that has been previously irradiated.
5. Prior anti-CTLA4 or anti-PD1 immunotherapy.
6. Active human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
7. A positive test for hepatitis B virus surface antigen (HBsAg) or hepatitis C antibody (HCV Ab).
8. Subjects with any active autoimmune disease or a documented history of autoimmune disease, except for:

   * Subjects with vitiligo
   * Resolved childhood asthma/atopy
   * Residual hypothyroidism due to an autoimmune condition requiring only hormone replacement
   * Psoriasis not requiring systemic treatment
   * Any condition not expected to recur in the absence of an external trigger.
9. Underlying medical conditions that, in the investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity or AE.
10. A concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids;
11. Pregnant or nursing.
12. A history of allergy to study drug components and/or a history of severe hypersensitivity to any monoclonal antibody.
13. Use of other investigational drugs 30 days before study drug administration and 5 half times before study inclusion.
14. Use of prohibited medication at start of study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Histopathological response rate at standard of care | At time of standard of care at week 4
  The proportion of viable tumor cells left in the resected specimen, to neo-adjuvant nivolumab and nivolumab plus ipilimumab at time of SOC (surgery ± RT).

SECONDARY OUTCOMES:
Sensitivity and specificity of tumor biopsies, clinical photography, FDG-PET and (functional)MRI compared to the histopathological tumor response to neo-adjuvant immunotherapy | At time of standard of care at week 4
  Histopathological tumor response to neo-adjuvant immunotherapy as measured in the tumor resection specimen will be compared to the tumor response as measured via serial tumor biopsies, the tumor biopsy at time of surgery and imaging (clinical photography, FDG-PET and (f)MRI). Histopathologic response in the tumor biopsies will be defined similarly as histopathologic response in the resected specimen. Response at imaging studies will be measured as follows: Clinical photography via specific clinical observation criteria, FDG-PET via RECIST 1.1 criteria and % change in TLG or MTV and (f)MRI via RECIST 1.1
Numbers of participants without significant delay (>1 week) or cancelation of SOC surgery due to immune-related toxicity | At time of standard of care at week 4
Recurrence free survival (RFS) at 2 years FU of responders versus non-responders to neo-adjuvant ICI | At 2-years follow up
Overall survival (OS) at 2 years FU of responders versus non-responders to neo-adjuvant ICI | At 2-years follow up
The number of patients with AE (rate and type) acoording to NCI CTCAE v.5.0 up to 2 years FU after SOC | At 2-years follow up
Clinical response of potentially additional AK surface areas after ICI identified by digital clinical photography on day 0, day 14, day 28 and every 6 months during FU up to 2 years. | On day 0, day 14, day 28 (at time of surgery) and every 6 months during FU up to 2 years.
Quality of life as measured by EORTC QLQ-C30 | At baseline, at surgery (week 4) and after 3, 6, 9, 12, 18 and 24 months during FU
  Rated on a Likert-type scale from one (never) to four (almost always), to evaluate different domains. Functional and global health status scales indicated towards better levels of functioning, whereas higher scores in the symptom scales demonstrated higher levels of symptoms.
Quality of life as measured by H&N 35 | At baseline, at surgery (week 4) and after 3, 6, 9, 12, 18 and 24 months during FU
  Rated on a Likert-type scale from one (never) to four (almost always). Multi-item scales (pain, swallowing, senses, speech, social eating, social contact, and sexuality), and six symptom items (teeth problems, opening mouth, dry mouth, sticky saliva, coughing, and feeling ill). Higher scores in the symptom scales demonstrated higher levels of symptoms.
Quality of life as measured by the EQ5D, | At baseline, at surgery (week 4) and after 3, 6, 9, 12, 18 and 24 months during FU
  Domains: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. It also includes a VAS regarding patients' "Health Today" scored between 0 and 100. Each domain will be converted into categorical values (problems vs no problems).
Quality of life as measured by the cancer worry scale (CWS) | At baseline, at surgery (week 4) and after 3, 6, 9, 12, 18 and 24 months during FU
  Rated on a Likert-type scale from one (never) to four (almost always), which were summed to produce a total CWS score ranging from 8 to 32, with higher scores indicating more frequent worries about cancer.
Quality of life as measured by the IT questionnaire | At baseline, at surgery (week 4) and after 3, 6, 9, 12, 18 and 24 months during FU
  Rated on a Likert-type scale from one (never) to four (almost always), to evaluate toxicity after immunotherapy treatment.
Quality of life as measured by the sexuality questionnaire | At baseline, at surgery (week 4) and after 3, 6, 9, 12, 18 and 24 months during FU
  Rated on a Likert-type scale from one (never) to four (almost always), to evaluate problems in sexual functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Lotje Zuur, MD, PHD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- NKI-AVL, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data will not be transferred.

REFERENCES:
- [Derived] Breukers SE, Traets JJH, van Dijk SW, Ostos MM, Fraterman I, Crommelin RD, van der Hulst H, Qiao X, Boere T, van de Poll-Franse LV, Retel V, van der Noort V, Vos JL, Toppenberg AGL, van der Heijden M, Missale F, Balm F, van den Brekel M, Dirven R, Karakullukcu MB, Karssemakers L, Klop WMC, Lohuis PJFM, Schreuder WH, Smeele LE, van der Velden LA, Plasmeijer E, Smit LA, de Boer JP, Navran A, Westerink B, de Koekkoek-Doll PK, Castelijns J, Wondergem M, Vogel WV, Kuijpers A, van Houdt WJ, Onderwater S, Maas-Bannink E, Cornelissen S, Broeks A, Tijink BM, Devriese LA, de Bree R, Blank CU, Schumacher TN, Thommen DS, Haanen JBAG, Zuur CL. Neoadjuvant ipilimumab and nivolumab in resectable cutaneous squamous cell carcinoma: a randomized phase 2 trial. Nat Med. 2025 Dec;31(12):4055-4064. doi: 10.1038/s41591-025-03943-w. Epub 2025 Oct 8. PMID 41062829